CLINICAL TRIAL: NCT05542121
Title: Rehabilitation Using Community-Based Affordable Robotic Exercise Systems (Rehab CARES)
Brief Title: Rehab CARES In USA: Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Recupero Robotics LLC (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Mercy Living Independently for Elders (LIFE) - West Philadelphia (Trinity Health Pace) (Unknown); enAble Games LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 853607; R42HD104325 (NIH)
Record Dates: First submitted 2022-09-06; First posted 2022-09-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Placebo Comparator): 60 min OT sessions; 3 sessions per week; for 4 weeks;-- augmented Standard therapy - consisting of PT, OT and SLP. Clinical Assessment (B1-pre, B2-post, B3-follow-up#1, B4-follow-up#2).
  Interventions: Other: Standard of Care
- Robot-Assisted Therapy with Rehab CARES system (Experimental): 60 min sessions; 3 sessions per week; for 4 weeks;----of Upper Limb therapy using 1 or more affordable robots. Robot sessions can be group play and/or single play.
  Robot Assessment (B1-pre, B2-post, B3-follow-up#1, B4-follow-up#2)
  Interventions: Device: Robot-Assisted Therapy with Rehab CARES system

INTERVENTIONS:
Device: Robot-Assisted Therapy with Rehab CARES system — 60 min sessions; 3 sessions per week; for 4 weeks; Patients uses 1 or more affordable robots to exercise the UL with adaptive games assessments as OT; standard of care PT and SLP; Subjects' motor and cognitive impairment will be used to set the game and modes. The game parameters will be adjusted according to motor and cognitive impairment of that station's user while the controller will automatically adjust assisting or resisting torques experienced. The 60 minutes will be broken up into 15-minute training intervals.
  Arms: Robot-Assisted Therapy with Rehab CARES system
Other: Standard of Care — 60 min sessions; 3 sessions per week; for 4 weeks of OT, PT, and SLP
  Arms: Standard of Care

SUMMARY:
In Phase 2, Patients in a community-based setting who have had a stroke will be evaluated by rehabilitation professionals and asked to perform a battery of clinical assessments before and after standard of care and robot assisted therapy with Rehab CARES system of simple force-feedback robots that are adapted to deliver single and group therapy.

DETAILED DESCRIPTION:
In Phase 2, we will develop the hardware to allow three haptic robots to dock (a gym) and be configured to allow patients to play therapy games alone or collaboratively. We will test the safety and feasibility of the gym in a community-based rehabilitation setting. We will treat 36 patients randomized to either a control group getting standard of care therapy and a robot group receiving standard of care with upper limb therapy being given using the robot gym instead of an occupational therapist. Therapy will occur over 4 weeks with two follow-up assessments. Key milestones will be to show that the robot group has the same or better functional outcomes, motivation, and adverse events as the control group. Also to show that the robot gym is a cost-effective solution to increasing access to quality rehabilitation care in low-resource, community-based settings. Success here will validate this potential solution, justify design changes revealed via user-feedback and a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 and older (based on who is admitted to the CBR site)
* >3 months post-stroke
* Stroke diagnosis
* Diagnosis of hemiparesis as a result of stroke (verified by radiology data)
* Motor control score on Upper Extremity Fugl-Meyer scale > 15 and < 60;
* Able to understand and speak
* Upper arm manual muscle strength scores >1
* Pain Scores < 8 based on NIH Pain Intensity Scale

Exclusion Criteria:

* no cerebellum lesions due to stroke
* severe cognitive function

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Motor Control | After 12 sessions (post-pre), after follow-up at 4 weeks (post-follow-up)
  Measured by Change in Upper Extremity Fugl-Meyer Assessment (UE-FM); scale is out of 66. A lower score means more impaired.
Change in Gross Hand Function | After 12 sessions (post-pre), after follow-up at 4 weeks (post-follow-up)
  Measured by Changes in Box and Block (BnB) Test; metric # of blocks transferred. A higher score means less impaired.
Change in Hand Dexterity | After 12 sessions (post-pre), after follow-up at 4 weeks (post-follow-up)
  Measured by changes in NIH Toolbox 9-Hole Pegboard Dexterity Test; metric time and # of peg transferred over time. A higher number of pegs means less impaired.
Upper Extremity Function | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by changes in the Neuro-QoL: Upper Extremity Function - Fine Motor, ADL Short Form. Short form is a self-report on 8 items to assesses fine motor function and activity of daily living in upper arm.
Quality of life (Participation) | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by changes in the Neuro-QoL: Ability to Participate in Social Role and Activities Short Form.
Quality of life (Satisfaction) | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by changes in Neuro-QoL Satisfaction with Social Roles and Activities Short Form.
Motivation | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by the Self-Assessment Manikin (SAM) scale which consist of 3 subscales: enjoyment, engagement, and control. Each subscale is from 0 to 9. For enjoyment and engagement the higher score is the better and for control the lower score is better.

SECONDARY OUTCOMES:
Change in Cognition | After 12 sessions (post-pre), after follow-up at 4 weeks (post-follow-up)
  Measured by changes in Montreal Cognitive Assessment (MocA)
Visual Spatial Attention | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by changes in Color Trails 1.A timed trail making assessment. A faster time result is better. Timed results are normalized by age and education and reported as a normalized z-score.
Executive Function | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by performance on Color Trails 2. A timed trail making assessment. A lower time is better. Timed results are normalized by age and education and reported as a normalized z-score.
Active Joint Range of Motion (ROM) | at pre, at post-intervention (after 12 sessions), at follow-up
  Range of Motion joint testing of the upper limb. Subjects shoulder, elbow, and wrist joint active joint movements are evaluated in the impaired arm. Reported in degrees.
Passive Joint Range of Motion (ROM) | at pre, at post-intervention (after 12 sessions), at follow-up
  Range of Motion joint testing of the upper limb. Subjects shoulder, elbow, and wrist joint passive joint movements are evaluated in the impaired arm. Reported in degrees.
Grip Strength | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by NIH toolbox Grip Strength Test. The amount of pound-force is measured. The higher pound-force is better.
Exertion Level | at each of 12 therapy sessions
  Measured by score on Borg Exertion Scale. Score is from 0 to 10. 0 is low and 10 is max. Subjects are asked to report pain experienced during a 60 minute session. Exertion between 0 and 6 is expected.
Pain Level | at each of 12 therapy sessions
  Measured by score on Visual Analog Pain Scale. Patients indicate a pain score is from 0 to 10. 0 is low and 10 is max. Subjects are asked to report pain experienced during a 60 minute session. Pain < 4 is expected.
Usability | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by score on System Usability Scale. Score is from 0 to 100. 0 is low and 100 is max. A score greater than or equal to 68 is ideal.
Work Load | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by NASA TLX Task Demand Scale. The scale consist of 6 questions scored on a likert scale of 0 to 21. The responses are processed to define a workload score. A workload score at or above 37 which is MOD-HIGH is expected.
Prediction of Motor Function | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by R-squared value from regression models of robot metrics from custom assessment tasks with respect to motor measurements of grip strength, gross hand function and fine motor function
Prediction of Cognitive Function | at pre, at post-intervention (after 12 sessions), at follow-up
  Measured by R-squared value from regression models of robot metrics from custom assessment tasks with respect to cognitive measurements of overall cognition, attention and executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle J Johnson, PhD, Principal Investigator — University of Pennsylvania; Alwyn Johnson, MS, Principal Investigator — Recupero Robotics LLC
Locations (2):
- United States (2):
  - Mercy Living Independently for Elders (L.I.F.E) - West Philadelphia, Philadelphia, Pennsylvania
  - Penn Medicine Rittenhouse, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
It is a priority of the research team to share primary data collected as a result of this project with other researchers and the National Institute of Health and associated funding agents. Findings will be disseminated within a reasonable time via newsletters sponsored by the institutions involved, peer-reviewed conference papers and journals. All journal papers will be placed on PubMed and made publically accessible. All acknowledgements will clearly define the funding agency and follow guidelines stipulated by the NIH. Copies of all publications will provided promptly. All copyright procedures will comply with the standard of NIH copyright clause.
  After study completion, de-identified data sets will be available to NIH and to other investigators contingent on the execution of relevant institutional data use agreements.
Supporting Information: Study Protocol, ICF
Time Frame: Within 2 years of project end
Access Criteria: Those wishing to see protocol and ICF will need to contact study PI